CLINICAL TRIAL: NCT05733819
Title: Responders to Metronome-based Rhythmic Auditory Cueing in Parkinson Disease
Brief Title: Responders to Rhythmic Auditory Cueing in Parkinson Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Terry Ellis, PT, PhD (Unknown)
Responsible Party: Principal Investigator, Lou Awad, PT, DPT, PhD, Assistant Professor, Boston University Charles River Campus
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 4440-PD
Record Dates: First submitted 2023-01-31; First posted 2023-02-17 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
Keywords: rhythmic auditory stimulation (RAS); gait analysis
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Subjects will complete a 6MWT without RAS and then complete a 6MWT with RAS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walking without personalized rhythmic auditory stimulation (Active Comparator): Subjects will complete a 6MWT without any auditory cues
  Interventions: Behavioral: Active Walking
- Walking with personalized rhythmic auditory stimulation (Experimental): Subjects will complete a 6MWT with personalized rhythmic auditory cues
  Interventions: Device: Subject-specific optimized RAS; Behavioral: Active Walking

INTERVENTIONS:
Device: Subject-specific optimized RAS — Walking with metronome-based RAS cueing
  Other Names: RAS
  Arms: Walking with personalized rhythmic auditory stimulation
Behavioral: Active Walking — Walking without RAS cueing

SUMMARY:
Parkinson disease (PD) is the second most common neurodegenerative disease affecting approximately 10 million people worldwide. It is a complex movement disorder that results in reduced walking ability. Prior studies have identified declines in walking as a marker of ensuing disability. Rhythmic auditory stimulation (RAS) is a rehabilitation approach that employs the coupling of auditory cues with movement. Walking with RAS has been shown to benefit walking rhythmicity, quality, and speed. These walking benefits make RAS advantageous in promoting regular moderate-intensity walking activity -- an important health objective in the management of PD. However, there is limited research investigating the effects of RAS on walking quality and how improvements in walking speed are achieved. This study will enroll 30 individuals with mild to moderate PD where each participant will be asked to complete two six-minute walk tests, one standard test (baseline) and the other using an optimized metronome-based auditory cueing RAS intervention. The investigators hypothesize that individuals with PD will either walk farther or with more automaticity (i.e., reduced stride time variability) in the RAS condition compared to the baseline condition. Moreover, these walking improvements will be accompanied by improvements in gait mechanics and metabolic cost of walking.

DETAILED DESCRIPTION:
Parkinson Disease (PD) is one of the fastest-growing sources of disability among neurological populations. PD is a progressive movement disorder characterized by substantial walking-related disability. Loss of function and quality of walking can subsequently lead to declines in walking which can precipitate a cycle of disability and deconditioning. In particular, persons with PD often demonstrate a reduction in stride length and an increase in stride time variability. These gait changes can reduce mobility and increase the risk of falls. Improving walking has been identified as the greatest priority among persons with PD for improving independence and quality of life. Therefore, interventions targeting improvements in walking function and gait quality are needed to mitigate a walking-related disability.

Rhythmic Auditory Stimulation (RAS) is a rehabilitation intervention that, unlike pharmacologic treatment, has shown promise for improving walking in PD. Walking with RAS intervention has been shown to improve walking function, particularly walking speed. RAS relies on the robust human capacity to synchronize movements to an external rhythm (i.e., walking to a regular auditory beat), a process referred to as auditory-motor entrainment. Due to the body's preference to select a walking frequency that maximizes stability and minimizes energy expenditure, rhythmic entrainment may stabilize gait patterns and reduce the metabolic cost of walking. Moreover, rhythmic entrainment is thought to reduce the attentional demand of walking in persons with PD, allowing for attention to be allocated to secondary tasks essential for safe community navigation. Despite evidence of the effectiveness of improving walking speed and gait function, the biomechanical changes that enable this improvement are not well understood.

Moreover, while RAS is an effective treatment, not everyone benefits from the treatment equally. Individuals with PD have a wide variety of gait presentations, and gait impairment may affect the efficacy of RAS treatment. In this study, the investigators want to understand who responds to RAS interventions and if the investigators can identify these responders from baseline measurements. For this analysis, the investigators define responders in three ways: (1) individuals who increase walking function, (2) individuals who increase gait quality, or (3) individuals who increase both gait quality and walking function while walking to personalized RAS. The investigators hypothesize that individuals who increase walking function and/or gait quality while walking to personalized RAS are more likely to be responsive to long-term intervention with RAS; however, the mechanism of action that enables the long-term response is hypothesized to be different based on baseline deficits. The investigators posit that the short-term responses to RAS measured in this study may suggest potential long-term mechanisms.

Study Protocol:

To examine the different effects of the intervention, each participant will complete a data collection session with a series of clinical tests including the Mini-BEST, UPDRS, the 10-m walk test (10MWT) at comfortable and fast walking speed, and the 6-minute walk test (6MWT) to quantity baseline function. Moreover, the 6MWT will be fully instrumented using motion capture cameras that track retro-reflective markers, wireless inertial measurement units, and force plates embedded in the walkway---together, these systems will enable concurrent collection of gait kinematic, inertial, and kinetic signals respectively. Additionally, metabolic measures will be collected during the 6MWT. After the baseline 6-minute walk test, participants will wear a custom, simple RAS device that will use a metronome application and bone-conducting headphones to provide auditory cues designed to modulate the participant's walking cadence. The auditory cues provided will be subject-specific based on a tuning procedure. Finally, the 6MWT will be repeated with RAS set to the optimally selected cadence based on the tuning procedure.

The primary objective of this study is to determine the effect of personalized RAS on walking function (i.e., 6MWT total distance) and gait quality (i.e., stride time variability). The investigators will also evaluate RAS-induced changes in other, secondary gait quality metrics: (1) the metabolic cost of transport, (2) walking ground reaction forces, (3) joint kinetics, and (4) distance-induced changes in spatial-temporal gait parameters. A secondary objective is to determine if RAS-induced changes in walking function and/or gait quality are related to specific patterns of baseline walking and gait impairment (i.e., movement phenotypes).

ELIGIBILITY:
Inclusion Criteria:

* Be able to communicate with investigators clearly
* Diagnosis of Parkinson's disease (self-report)
* The ability to walk continuously without another individual supporting the person's body weight for at least 6 minutes. Assistive devices, such as a cane, are allowed.

Exclusion Criteria:

* Inability to communicate (as assessed by a licensed physical therapist)
* Parkinson's disease, score < 23 on the MMSE.
* Pain that impairs walking ability (as assessed by a licensed physical therapist)
* Unexplained dizziness in the last 6 months (self-report)
* Severe comorbidities that may interfere with the ability to participate (musculoskeletal, cardiovascular, pulmonary, and neurological)
* More than 2 falls in the previous month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Six Minute Walk test distance | [RAS-Baseline]
  difference in total distance walked with and without RAS. (m)
Stride time variability | [RAS-Baseline]
  difference in stride time variability with and without RAS (%)

SECONDARY OUTCOMES:
Metabolic Cost of Transport | [RAS-Baseline]
  difference in energy cost of walking with and without RAS. Metabolic cost of transport is defined as metabolic energy (measured directly from COSMED) per kg of body weight (in mL/s/kg or W/kg) divided by the average speed during the six minute walk test (mL/kg/m or J/kg/m).
Ground Reaction Forces | [RAS-Baseline]
  difference in Anterior Posterior GRF -- including both peak and impulse (%bw)
Joint power | [RAS-Baseline]
  difference in joint power computed using inverse dynamics -- including ankle, knee, and hip moment. (W/kg)
speed changes over the 6MWT | [RAS-Baseline]
  the difference in changes in walking speed over the 6MWT (m/s)
stride length changes over the 6MWT | [RAS-Baseline]
  the difference in changes in stride length over the 6MWT (cm)
cadence changes over the 6MWT | [RAS-Baseline]
  the difference in changes in cadence over the 6MWT (steps/min)

OTHER OUTCOMES:
Joint moments | [RAS-Baseline]
  difference in joint moments computed using inverse dynamics -- including ankle, knee, and hip moment. (Nm/kg)
spatial temporal relationships over the 6MWT | [RAS-Baseline]
  difference in changes in relationship (linear regression) between speed: cadence, speed: stride length and cadence: stride-length

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University Neuromotor Recovery Laboratory, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified subject data with and without RAS may be published as part of the manuscript. Data may include, kinematics, kinetics, metabolic and clinical data.
Time Frame: At the time of manuscript acceptance

REFERENCES:
- [Background] Shulman LM, Gruber-Baldini AL, Anderson KE, Vaughan CG, Reich SG, Fishman PS, Weiner WJ. The evolution of disability in Parkinson disease. Mov Disord. 2008 Apr 30;23(6):790-6. doi: 10.1002/mds.21879. PMID 18361474
- [Background] Shulman LM. Understanding disability in Parkinson's disease. Mov Disord. 2010;25 Suppl 1:S131-5. doi: 10.1002/mds.22789. PMID 20187231
- [Background] Lord S, Godfrey A, Galna B, Mhiripiri D, Burn D, Rochester L. Ambulatory activity in incident Parkinson's: more than meets the eye? J Neurol. 2013 Dec;260(12):2964-72. doi: 10.1007/s00415-013-7037-5. Epub 2013 Jul 31. PMID 23900754
- [Background] Cavanaugh JT, Ellis TD, Earhart GM, Ford MP, Foreman KB, Dibble LE. Capturing ambulatory activity decline in Parkinson's disease. J Neurol Phys Ther. 2012 Jun;36(2):51-7. doi: 10.1097/NPT.0b013e318254ba7a. PMID 22592060
- [Background] Cochen De Cock V, Dotov D, Damm L, Lacombe S, Ihalainen P, Picot MC, Galtier F, Lebrun C, Giordano A, Driss V, Geny C, Garzo A, Hernandez E, Van Dyck E, Leman M, Villing R, Bardy BG, Dalla Bella S. BeatWalk: Personalized Music-Based Gait Rehabilitation in Parkinson's Disease. Front Psychol. 2021 Apr 26;12:655121. doi: 10.3389/fpsyg.2021.655121. eCollection 2021. PMID 33981279
- [Background] Forte R, Tocci N, De Vito G. The Impact of Exercise Intervention with Rhythmic Auditory Stimulation to Improve Gait and Mobility in Parkinson Disease: An Umbrella Review. Brain Sci. 2021 May 22;11(6):685. doi: 10.3390/brainsci11060685. PMID 34067458
- [Background] Nonnekes J, Nieuwboer A. Towards Personalized Rehabilitation for Gait Impairments in Parkinson's Disease. J Parkinsons Dis. 2018;8(s1):S101-S106. doi: 10.3233/JPD-181464. PMID 30584154
- [Background] Port RJ, Rumsby M, Brown G, Harrison IF, Amjad A, Bale CJ. People with Parkinson's Disease: What Symptoms Do They Most Want to Improve and How Does This Change with Disease Duration? J Parkinsons Dis. 2021;11(2):715-724. doi: 10.3233/JPD-202346. PMID 33459664
- [Background] Burrai F, Apuzzo L, Zanotti R. Effectiveness of Rhythmic Auditory Stimulation on Gait in Parkinson Disease: A Systematic Review and Meta-analysis. Holist Nurs Pract. 2024 Mar-Apr 01;38(2):109-119. doi: 10.1097/HNP.0000000000000462. Epub 2021 Jun 11. PMID 34121062
- [Background] Ye X, Li L, He R, Jia Y, Poon W. Rhythmic auditory stimulation promotes gait recovery in Parkinson's patients: A systematic review and meta-analysis. Front Neurol. 2022 Jul 28;13:940419. doi: 10.3389/fneur.2022.940419. eCollection 2022. PMID 35968291
- [Background] Erra C, Mileti I, Germanotta M, Petracca M, Imbimbo I, De Biase A, Rossi S, Ricciardi D, Pacilli A, Di Sipio E, Palermo E, Bentivoglio AR, Padua L. Immediate effects of rhythmic auditory stimulation on gait kinematics in Parkinson's disease ON/OFF medication. Clin Neurophysiol. 2019 Oct;130(10):1789-1797. doi: 10.1016/j.clinph.2019.07.013. Epub 2019 Jul 25. PMID 31401487
- [Background] Nombela C, Hughes LE, Owen AM, Grahn JA. Into the groove: can rhythm influence Parkinson's disease? Neurosci Biobehav Rev. 2013 Dec;37(10 Pt 2):2564-70. doi: 10.1016/j.neubiorev.2013.08.003. Epub 2013 Sep 3. PMID 24012774
- [Background] Ashoori A, Eagleman DM, Jankovic J. Effects of Auditory Rhythm and Music on Gait Disturbances in Parkinson's Disease. Front Neurol. 2015 Nov 11;6:234. doi: 10.3389/fneur.2015.00234. eCollection 2015. PMID 26617566